CLINICAL TRIAL: NCT02193061
Title: Randomized, Controlled Single-blind Clinical Study to Assess Vaccine Interchangeability Between Rota Vaccine 5 and Rota Vaccine 1 Using Seven Combined Anti-rotavirus Prevention Programs: ROTA 1,ROTA 2,ROTA 3,ROTA 4,ROTA 5,ROTA 6,ROTA 7 in Infants at 2, 4 and 6 Months of Age in Mexico City.
Brief Title: Randomized, Controlled Single-blind Clinical Study to Assess Vaccine Interchangeability Between RV5 and RV1 Using Seven Combined Anti-rotavirus Prevention Programs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Pediatrics, Mexico (Other Government)
Collaborators: Centro Nacional para la Salud de la Infancia y la Adolescencia (Other Government); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Mercedes Macias Parra, MSc, National Institute of Pediatrics, Mexico
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Rota/CeNSIA
Record Dates: First submitted 2014-07-07; First posted 2014-07-17 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Rotavirus Vaccine
Keywords: Rotavirus; immunological behavior; Rotarix; RotaTeq; vaccine interchangeability
MeSH Terms: interventions — RIX4414 vaccine; RotaTeq

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- ROTA 1 (Active Comparator): two doses of monovalent vaccine Rotarix followed by one dose of sterile water
  Interventions: Biological: Rotarix
- ROTA 2 (Active Comparator): three doses of pentavalent vaccine RotaTeq
  Interventions: Biological: RotaTeq
- ROTA 3 (Active Comparator): one dose of monovalent Rotarix vaccine followed by two doses of pentavalent vaccine Rotateq
  Interventions: Biological: Rotarix; Biological: RotaTeq
- ROTA 4 (Active Comparator): one dose of pentavalent RotaTeq vaccine followed by two doses of monovalent vaccine Rotarix
  Interventions: Biological: Rotarix; Biological: RotaTeq
- ROTA 5 (Active Comparator): two doses of pentavalent vaccine RotaTeq followed by a dose of monovalent vaccine Rotarix
  Interventions: Biological: Rotarix; Biological: RotaTeq
- ROTA 6 (Active Comparator): one dose of pentavalent vaccine RotaTeq followed by a dose of monovalent vaccine Rotarix and a dose of pentavalent vaccine RotaTeq
  Interventions: Biological: Rotarix; Biological: RotaTeq
- ROTA 7 (Active Comparator): a dose of monovalent vaccine Rotarix followed by a dose of pentavalent vaccine and a dose of monovalent vaccine Rotarix
  Interventions: Biological: Rotarix; Biological: RotaTeq

INTERVENTIONS:
Biological: Rotarix
  Arms: ROTA 1; ROTA 3; ROTA 4; ROTA 5; ROTA 6; ROTA 7
Biological: RotaTeq
  Arms: ROTA 2; ROTA 3; ROTA 4; ROTA 5; ROTA 6; ROTA 7

SUMMARY:
Assess the immunological behavior of children from 2 months of age that receive one out of seven anti-rotavirus vaccination programs: Group 1 (routine schedule with two doses of RV1 - Rotarix plus sterile water) and Group 2 (routine schedule with three doses of RV5 - RotaTeq) versus Group 3 (one dose of monovalent vaccine followed by two doses of pentavalent vaccine), Group 4 (one dose of pentavalent vaccine followed by two doses of monovalent vaccine), Group 5 (two doses of pentavalent vaccine followed by a dose of monovalent vaccine), Group 6 (one dose of pentavalent vaccine followed by a dose of monovalent vaccine and a dose of pentavalent vaccine), and Group 7 (a dose of monovalent vaccine followed by a dose of pentavalent vaccine and a dose of monovalent vaccine) in children from Mexico City.

Secondary objectives

* To describe number and features of acute diarrheal disease (ADD) due to rotavirus displayed in the seven prevention schedules.
* To describe the adverse events temporarily associated with the seven prevention schedules.

Hypotheses The seroconversion percentages and geometric mean titers (GMT) of anti-rotavirus antibodies from Groups 3, 4, 5, 6 and 7 are not inferior to the seroconversion percentages and the GMTs induced in subjects that received the routine vaccination schedules with two doses of the monovalent vaccine and three doses of the pentavalent vaccine (Groups 1 and 2).

DETAILED DESCRIPTION:
In this protocol we included 1498 at 6 to 8 weeks of age with a second visit at 2 months, a third visit at 4months four visit at 5 months after the first vaccination, ( 1st, second and 3erd visits for vaccine administration) phone calls every month and not schedule visits at the center when parents required and the last protocol visit was at one year of age This follow up to one year was to access security.

ELIGIBILITY:
Inclusion Criteria:

* The subject is a boy or a girl 2 months ± one week old at the time of the first dose of the vaccine.
* The subject is considered to be healthy based on the clinical history and the physical examination.
* The subject has not received any anti-rotavirus vaccine.
* The parent/tutor fully understands the study's procedures and voluntarily accepts to participate and signs a written informed consent.
* The parent/tutor can meet the study's requirements, such as attending the programmed visits and filling in the journal.
* Written informed consent signed by the parent/tutor before any procedure.

Exclusion Criteria:

* The subject has a background of serious allergic reaction to any of the vaccine's components.
* The subject has a digestive tract malformation or acute/chronic disease.
* The subject has some kind of immunodeficiency including HIV.
* The subject suffers from a haemato-oncological disease.
* The subject has been under treatment with an immunosuppressing medicine including prednisone for two or more weeks.
* The subject has received gamma-globulin or any other blood-derived product or its administration is programmed during the study.

Ages: 6 Weeks to 10 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1498 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
General Symptoms - Temperature | subsequent 5 days since the vaccination day
  The subject temperature will be registered with a rectal thermometer during 5 days since the vaccination day in a diary card .
  If the subject presents fever, the temperature will be recorded in a specific diary card section.

SECONDARY OUTCOMES:
Evacuation | subsequent 30 days since the vaccination day
  The number of evacuations per day and their characteristics will be registered in a diary card

CONTACTS AND LOCATIONS:
Locations (1):
- National Instiute of Pediatrics, México, D.F., Mexico

REFERENCES:
- [Derived] Macias-Parra M, Vidal-Vazquez P, Reyna-Figueroa J, Rodriguez-Weber MA, Moreno-Macias H, Hernandez-Benavides I, Fortes-Gutierrez S, Richardson VL, Vazquez-Cardenas P. Immunogenicity of RV1 and RV5 vaccines administered in standard and interchangeable mixed schedules: a randomized, double-blind, non-inferiority clinical trial in Mexican infants. Front Public Health. 2024 Feb 23;12:1356932. doi: 10.3389/fpubh.2024.1356932. eCollection 2024. PMID 38463163